CLINICAL TRIAL: NCT01953822
Title: An Observational Cohort Study to Assess the Risk of Autoimmune Diseases in Adolescent and Young Adult Women Aged 9 to 25 Years Exposed to Cervarix® in the United Kingdom
Brief Title: Study Assessing Risk of Autoimmune Diseases in Females (9 - 25 Years) Exposed to Cervarix® in United Kingdom
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 116239
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2016-12

CONDITIONS: Infections, Papillomavirus
Keywords: Observational; Cohort; Autoimmune disease; Cervarix®; Women aged 9 to 25 years; United Kingdom
MeSH Terms: conditions — Papillomavirus Infections; Autoimmune Diseases | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (4):
- Cervarix vaccinated (exposed) female cohort: Female subjects vaccinated with at least one dose of Cervarix® between the ages of 9 to 25 years.
  Interventions: Other: Data collection
- Unexposed historical female cohort: Unexposed female subjects identified from historical data, will be frequency matched for age and practice region identifier to the subjects included in the vaccinated (exposed) cohort.
  Interventions: Other: Data collection
- Unexposed concurrent male cohort: Male population is composed of 9- to 25-year-old male subjects not vaccinated with Cervarix®.
  Interventions: Other: Data collection
- Unexposed historical male cohort: Male population is composed of 9- to 25-year-old male subjects not vaccinated with Cervarix®. Comparison of the unexposed concurrent male cohort with the unexposed historical male cohort will be used as an internal control for changes over time in Clinical Practice Research Datalink (CPRD) GOLD in reporting New Onset of Autoimmune Diseases (NOAD). The male subjects will be frequency matched for age and practice region identifier to the subjects included in the vaccinated (exposed) cohort.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data collection from an existing electronic healthcare databases - Clinical Practice Research Datalink (CPRD) GOLD.

SUMMARY:
This is an observational cohort study to assess the risk of autoimmune disease(s) within 12 months of receiving the first dose of Cervarix® in the exposed cohort and over a comparable period in the unexposed cohorts.

This is an alternative study by GSK using the CPRD database in the UK to fulfil the US FDA safety commitment. The UK has had sufficient Cervarix® vaccination coverage during the period mid-September 2008 to 2011 to allow suitable data to be collected.

DETAILED DESCRIPTION:
GSK's vaccine Cervarix® protects against Human Papilloma Virus Types-16 and 18-related pre-cancerous lesions. GSK is committed by the US Food and Drug Administration (FDA) to conduct a safety study to evaluate the incidence of new neurological and eye-related autoimmune diseases and other pre-specified autoimmune diseases in subjects receiving Cervarix® in the US. Because of the very low Cervarix® uptake in the US, the observational GSK study to address this commitment is due to be stopped, as it will take too long to recruit the target subjects.

The unexposed male cohorts will be enrolled in order to assess a possible change over time in the incidence rate of new onset of autoimmune disease(s) (NOAD) in the UK Clinical Practice Research Datalink General Practitioner OnLine database (CPRD GOLD) independent of Cervarix® introduction. The cohorts will be frequency matched for the age (age class of one year) and practice region identifier at reference date (age at first dose of Cervarix).

Additionally, the reference date (time = 0) for the vaccinated (exposed) cohort will be the date of the first dose of Cervarix® recorded in CPRD GOLD. The reference date for the unexposed (unvaccinated) cohorts will be a date randomly selected among the reference dates of the exposed subjects and minus 3 years for the historical cohorts.

The other observational study model is a self-control case-series (SCCS) analysis for confirmed NOAD in the exposed female cohort, using a risk period of one year after the first Cervarix® dose, a control period of one year and a six month buffer period between risk and control periods.

Human Papillomavirus Bivalent (Types 16 and 18) vaccine (recombinant) exposed cohort was investigated between 1-SEP-2008 and 31-AUG-2010.

The unexposed concurrent male cohort was investigated between 1-SEP-2008 and 31-AUG-2010.

Unexposed historical female and male cohorts were investigated between 1-SEP-2005 and 31-AUG-2007.

ELIGIBILITY:
Inclusion Criteria:

Note: Other vaccines are allowed in this study regardless of the time of administration and the time interval between subsequent doses.

Inclusion criteria for the exposed female cohort:

* Female aged from 9 to 25 years at the reference date (01 September 2008 through 31 August 2010).
* Recorded in the CPRD GOLD for at least 12 months before the reference date.
* The first dose of Cervarix received between 01 September 2008 through 31 August 2010, Full date (day/month/year) of Cervarix vaccination(s) available.
* Subject defined as acceptable in CPRD GOLD.

Inclusion criteria for the unexposed historical female cohort:

* Female aged 9 to 25 years at the reference date (01 September 2005 through 31 August 2007).
* Recorded in the CPRD GOLD for at least 12 months before the reference date.
* Subject defined as acceptable in CPRD GOLD.

Inclusion criteria for the unexposed concurrent male cohort:

* Male aged 9 to 25 years at the reference date (01 September 2008 through 31 August 2010).
* Recorded in the CPRD GOLD for at least 12 months before the reference date.
* Subject defined as acceptable in CPRD GOLD.

Inclusion criteria for the unexposed historical male cohort:

* Male aged 9 to 25 years at the reference date (01 September 2005 through 31 August 2007).
* Recorded in the CPRD GOLD for at least 12 months before the reference date.
* Subject defined as acceptable in CPRD GOLD.

Exclusion Criteria:

Exclusion criteria for all cohorts:

* Subjects with a diagnostic code of any auto-immune disease during the year prior to the reference date.
* Subjects who received at least one dose of unspecified HPV vaccine or Gardasil at any time before the reference date.
* Subjects who have been included in the other cohort.

Exclusion criteria for the non-exposed cohorts:

• Subjects who received any dose of Cervarix at any time before the reference date.

Ages: 9 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Female population is composed of female subjects vaccinated with Cervarix® between the ages of 9 to 25 years and unexposed female subjects identified from historical data. Male population is composed of 9- to 25-year-old male subjects not vaccinated with Cervarix®.
Sampling Method: Non-Probability Sample
Enrollment: 1053 (Actual)
Dates: Start 2013-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Occurrence of new onset of confirmed autoimmune disease for neuroinflammatory/ophthalmic autoimmune diseases | During the period of 1 year following administration of the first dose of Cervarix® (risk period) among an exposed cohort and during an equivalent time period in the unexposed cohorts
  Neuroinflammatory/ophthalmic autoimmune diseases: -Multiple Sclerosis; -Transverse myelitis; -Optic neuritis; -Guillain-Barré syndrome, including Miller Fisher syndrome and other variants; -Other demyelinating diseases: -Acute disseminated encephalomyelitis, including site specific variants: e.g. non-infectious encephalitis, encephalomyelitis, myelitis, myeloradiculomyelitis; -AI peripheral neuropathies and plexopathies (including chronic inflammatory demyelinating polyneuropathy, multifocal motor neuropathy and polyneuropathies associated with monoclonalgammopathy); -Auto-immune uveitis;
Occurrence of new onset of confirmed autoimmune disease for other autoimmune diseases | During the period of 1 year following administration of the first dose of Cervarix® (risk period) among an exposed cohort and during an equivalent time period in the unexposed cohorts
  Other autoimmune diseases: -Systemic lupus erythematous; -Autoimmune (AI) disease with rheumatologic conditions: -Rheumatoid arthritis (RA);-Juvenile rheumatoid arthritis (JRA); -Still's disease; -Psoriatic arthritis; -Ankylosing Spondylitis; -AI haematological conditions: -Idiopathic thrombocytopenic purpura (ITP); -AI haemolytic anaemia; -AI endocrine conditions: -Type 1 diabetes mellitus; -AI thyroiditis including Hashimoto's disease, Graves' /Basedows' disease; -Inflammatory bowel / hepatic diseases: -Crohn's diseases; -Ulcerative colitis; -Autoimmune hepatitis;

SECONDARY OUTCOMES:
Occurrence of Guillain Barré syndrome (including Miller Fisher syndrome and other variants), and autoimmune haemolytic anaemia | Within 2 months following the administration of the first dose of Cervarix®
Occurrence of idiopathic thrombocytopenic purpura (ITP) | Within six months following the administration of the first dose of Cervarix®
Occurrence of new onset of individual confirmed autoimmune disease | Within 1 year following the administration of the first dose of Cervarix®
  Occurrence of multiple sclerosis, transverse myelitis, optic neuritis, other demyelinating diseases, auto-immune uveitis, systemic lupus erythematous (SLE), rheumatoid arthritis (RA), juvenile rheumatoid arthritis (JRA), Still's disease, psoriatic arthritis, ankylosing spondylitis, type 1 diabetes mellitus, auto-immune thyroiditis (including Hashimoto's disease, Graves'/Basedows' disease), and inflammatory bowel / hepatic disease (Crohn's disease, ulcerative colitis and autoimmune hepatitis)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline